CLINICAL TRIAL: NCT01489696
Title: A Study to Evaluate Cardiovascular Interactions Between Mirabegron and Tamsulosin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 178-CL-080; 2010-018690-38 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-12-12 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Cardiovascular; Healthy Subjects; Pharmacokinetics
Keywords: Pharmacokinetics; Mirabegron; Tamsulosin; Phase 1
MeSH Terms: interventions — mirabegron; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm 1 (Experimental): tamsulosin singles doses; mirabegron multiple dose
  Interventions: Drug: mirabegron; Drug: tamsulosin
- Treatment Arm 2 (Experimental): mirabegron single doses; tamsulosin multiple dose
  Interventions: Drug: mirabegron; Drug: tamsulosin

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178
Drug: tamsulosin — oral
  Other Names: Flomax; Harnal; Omnic

SUMMARY:
The study aims to compare blood pressure and pulse in male healthy subjects taking mirabegron and tamsulosin both alone and in combination.

DETAILED DESCRIPTION:
Treatment arm 1 (effect of mirabegron on tamsulosin): Subjects are randomized into one of two sequences.

Subjects receive 2 singles doses of tamsulosin, once in the absence of mirabegron and once in the presence of mirabegron.

24-hour Cardiovascular (CV) profiles are taken at both baseline days and after the single dose of tamsulosin /combination dose in each sequence. Regular blood samples are also taken to check for a potential Pharmacokinetic (PK) interaction.

Treatment arm 2 (effect of tamsulosin on mirabegron): Subjects are randomized into one of two sequences.

Subjects receive 2 singles doses of mirabegron, once in the absence of tamsulosin and once in the presence of tamsulosin.

24-hour CV profiles are taken at both baseline days and after the single dose of mirabegron/combination dose in each sequence. Regular blood samples are also taken to check for a potential PK interaction.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index more than or equal to 18.5 and less than 30.0 kg/m2

Exclusion Criteria:

* Known or suspected hypersensitivity to mirabegron and/or tamsulosin HCl, or any components of the formulations used
* Any of the liver function tests (i.e. Alanine Aminotransferase (ALT) and Asparate Aminotransferase (AST) above the upper limit of normal at repeated measures (at least one more time)
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever)
* Any prior clinically significant psychiatric history including hospitalization for mental health management
* Subject is at risk of urinary retention based on medical history
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, Electrocardiogram (ECG) and clinical laboratory tests
* Heart rate and/or blood pressure measurements at the screening and admission visits as follows: Heart rate <50 or >90 bpm; mean systolic blood pressure <90 mm Hg or >140 mmHg (>160 mmHg for subjects 65 years or older); mean diastolic blood pressure <60 mm Hg or >90 mmHg (>100 mmHg for subjects 65 years or older) (blood pressure measurements to be taken after subject has been resting in supine position for 5 min; heart rate will be measured automatically; both to be taken in triplicate)
* A QTc interval of > 430 ms after repeated measurements (at least two more times), a history of syncope, orthostatic hypotension, vertigo, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)
* A hemoglobin value <12.5 g/dl (7.8 mmol/l) and/or a hematocrit value <37.9% and/or a Red Blood Cell count <4.08 T/l (4080 mm3)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular interactions assessed by blood pressure and pulse rate | Pre-dose until 24 hours after dosing

SECONDARY OUTCOMES:
Monitoring of safety and tolerability through assessment of vital signs, ECG, clinical safety laboratory and adverse events | Arm 1: From time of combination dose until 4 days after combination dose / Arm 2: From time of combination dose until 8 days after combination dose
Potential PK interaction of the combination dosing assessed by serial plasma sampling | Arm 1: From time of combination dose until 4 days after combination dose (10 time points) / Arm 2: From time of combination dose until 8 days after combination dose (14 time points)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Covance CRU Ltd, Leeds, United Kingdom